CLINICAL TRIAL: NCT01372566
Title: Effect of Autologous Platelet-rich Plasma on Photoaged Skin: A Prospective Randomized Controlled Trial (Phases A and B)
Brief Title: Effect of Platelet Rich Plasma on Photoaged Skin
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STU34547
Record Dates: First submitted 2011-06-01; First posted 2011-06-14 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Photoaging

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Rich Plasma (Experimental): Concentrated blood platelets from subject will be injected multiple times into the superficial layer of either their arm (Part 1) or one side of their upper face and cheek (Part 2).
  Interventions: Device: Harvest PRP Separation System
- Sterile Saline (Placebo Comparator): Sterile saline will be injected multiple times into the superficial layer of either their arm (Part 1) or one side of their upper face and cheek (Part 2)that has not been injected with PRP.
  Interventions: Other: Sterile Saline injection

INTERVENTIONS:
Device: Harvest PRP Separation System — Platelet-rich plasma (PRP) is a blood-derived therapy that consists of platelets and growth factors. PRP can be formed by drawing blood from a vein and spinning it at a high speed in a specialized device called a centrifuge.
  Arms: Platelet Rich Plasma
Other: Sterile Saline injection — Sterile Saline will be injected multiple times in a different area of the arm (Part 1) or on the opposite side of the face from where the platelet rich plasma is injected.
  Arms: Sterile Saline

SUMMARY:
The goal of this study is to assess the safety, tolerability and effectiveness of platelet rich plasma in the treatment of photoaged skin. This study will be divided into two parts. The first part will assess the safety and tolerability of platelet rich plasma injections as compared to sterile saline injections in subjects' arm with six months follow-up. The second part will assess the effect of platelet rich plasma on the appearance of facial skin in a split face study with platelet rich plasma injections on one side of the face and sterile saline on the other. Outcomes will be recorded for twelve months.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Subjects of either gender (M/F), 35-60 years old.
* Subjects are in good health.
* Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Part 2:

* Subjects of either gender (M/F), 35-60 years old.
* Subjects are in good health.
* Bilateral cheek wrinkles "in motion" with severities of ≥ type II of Glogau photoaging classification (APPENDIX I).
* Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.
* Subject requests cosmetic improvement of facial wrinkles.

Exclusion Criteria:

* Pregnant or lactating.
* Subjects who are unable to understand the protocol or to give informed consent.
* Subjects who have a self-reported history of blood or platelet disorders e.g. anemia, thrombocytopenia, coagulopathy, hypofibrinogenemia, or are on anticoagulant or antiplatelet therapy.
* Subjects who have active skin disease or skin infection in treatment area. Subjects who have a history of hypertrophic scars and keloids.
* Subjects who have any requirement for the use of local or systemic steroids or immunosuppressive agents.
* Subject notes that he/she is HIV positive
* Subjects with history of skin cancer or actinic keratosis
* Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
* Skin conditions that interfere with wrinkle assessment/treatment (excessive dermatochalasis, inability to lessen the wrinkles by physically spreading the area apart).
* Excessive exposure to the sun, such as jobs requiring constant outdoor exposure.
* Known genetic disorders affecting fibroblasts or collagen, such as achondroplasia, osteogenesis imperfecta, ect.

Part 2:

* Pregnant or lactating.
* Subjects who are unable to understand the protocol or to give informed consent.
* Subjects who have a history of blood or platelet disorders e.g. anemia, thrombocytopenia, coagulopathy, hypofibrinogenemia, or are on anticoagulant or anti-platelet therapy.
* Subjects who have had topical or oral tretinoin, chemical peeling, botulinum toxin injection or laser and light treatment for facial rhytides or rejuvenation within past 6 months or planning to undergo treatments as described in the next 3 months.
* Facial surgery in the lower 2/3 of the face or semi-permanent dermal fillers within 1 year prior to study enrollment
* Subjects who have history of recurrent facial or labial herpes simplex infection.
* Subjects who have active skin disease or skin infection in treatment area.
* Subjects who are allergic to lidocaine or prilocaine.
* Subjects who have a history of hypertrophic scars and keloids.
* Subjects who have any requirement for the use of local or systemic steroids or immunosuppressive agents.
* Subject notes that he/she is HIV positive
* Subjects with history of skin cancer or actinic keratosis
* Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
* Skin conditions that interfere with wrinkle assessment/treatment (excessive dermatochalasis, inability to lessen the wrinkles by physically spreading the area apart).
* Excessive exposure to the sun, such as jobs requiring constant outdoor exposure.
* Known genetic disorders affecting fibroblasts or collagen, such as achondroplasia, osteogenesis imperfecta, ect.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2011-05; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Study Part 1: Safety and Tolerability | 2 weeks, 1 month, 3 months and 6 months
  The primary outcome measures will be the evaluation of safety and tolerability, which will be assessed by collection of adverse events throughout the feasibility study.
Primary Outcome Study Part 2: Change in Photoaging scores from Baseline at 2 weeks, 3 months, and 6 months | Treatment visit, 2 weeks, 3 months and 6 months
  Photoaging scores will be recorded for each cheek by two blinded dermatologists at the treatment visit (before treatment)and during the 2 week, 3 month, and 6 month post-treatment visits. Individual scores for each variable (fine lines, mottled pigmentation, roughness, and sallowness) will be recorded by the blinded dermatologists.

SECONDARY OUTCOMES:
Secondary Outcome of Study Part 1: Histologic analysis | 1 month
  The secondary outcomes measures will involve the dermatopathologic review of the 2 skin biopsies taken from each subject at the one month post-treatment visit. One 3mm biopsy will be taken from the skin where the saline was injected and the other from the site of PRP injection. These will be reviewed by the dermatopathologists in the Department of Dermatology for significant histological changes, including collagen remodeling and possible reduction in photodamage. Histologic stains will include hematoxylin and eosin and Masson's trichrome.
Secondary Outcome Study Part 2: Self-Assessment | 3 and 6 months
  A subject self-assessment of each cheek will be performed at the 3 and 6 month follow up visits.
Secondary Outcome Study Part 2: Subject Satisfaction | 6 months
  A subject overall satisfaction questionnaire will be performed at the 6 month follow up visit.
Secondary Outcome Study Part 2: Rate of Adverse Events | 2 weeks, 3 months, 6 months, 12 months
  Adverse events will be recorded at each time point, if they occur. Statitical analysis will determine the rate of any adverse events between PRP and Saline.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Alam M, Hughart R, Champlain A, Geisler A, Paghdal K, Whiting D, Hammel JA, Maisel A, Rapcan MJ, West DP, Poon E. Effect of Platelet-Rich Plasma Injection for Rejuvenation of Photoaged Facial Skin: A Randomized Clinical Trial. JAMA Dermatol. 2018 Dec 1;154(12):1447-1452. doi: 10.1001/jamadermatol.2018.3977. PMID 30419125